CLINICAL TRIAL: NCT03731715
Title: Phase I, Open-Label, Pharmacokinetic, Dose Escalation Study of Carisbamate in Adult and Pediatric Subjects With Lennox-Gastaut Syndrome
Brief Title: Carisbamate in Adult & Pediatric Subjects With Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YKP509C001
Record Dates: First submitted 2018-10-16; First posted 2018-11-06 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Lennox Gastaut Syndrome
Keywords: LGS
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort I (Experimental): Subjects ≥18 years of age. Carisbamate, 200 mg, will be administered on Day 1 and 2 of the single-dose period. Carisbamate will be administered at 100 mg twice daily (BID) during the multiple-dose period.
  Interventions: Drug: Carisbamate
- Cohort II (Experimental): Subjects 12 to <18 years of age. Carisbamate, 140 mg, will be administered on Day 1 and 2 of the single dose period. Carisbamate will be administered at 70 mg twice daily (BID) during the multiple-dose period.
  Interventions: Drug: Carisbamate
- Cohort III (Experimental): Subjects 6 to <12 years of age. Carisbamate, 60 mg, will be administered on Day 1 and 2 of the single dose period. Carisbamate will be administered at 30 mg twice daily (BID) during the multiple-dose period.
  Interventions: Drug: Carisbamate
- Cohort IV (Experimental): Subjects 2 to <6 years of age. The starting doses for the single dose and multiple-dose periods will be based on the PK and safety results of the first 3 cohorts.
  Interventions: Drug: Carisbamate

INTERVENTIONS:
Drug: Carisbamate — An oral liquid formulation (20 mg/mL) of carisbamate (S-carisbamate)
  Other Names: YKP509

SUMMARY:
This is an open-label, multi-center study of carisbamate in adult and pediatric subjects with LGS, with single- and multiple-dose PK assessments from Days 1 through 73. There will be a Screening Period of up to 28 days and a Treatment Period of 87 days.

DETAILED DESCRIPTION:
A total of 24 subjects are planned: 6 subjects in each of 4 cohorts: Cohort I (≥18 years), Cohort II (12 to <18 years), Cohort III (6 to <12 years), and Cohort IV (2 to <6 years).

For Cohorts I and II, PK assessments of carisbamate, S-enantiomer and its R-enantiomer plasma concentrations, will be conducted on Days 1, 2 and 3 of the single dose period at pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 hours after dosing and on Day 17 of the multiple-dose period at pre dose and 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours after dosing; trough samples will be collected on Days 45 and 73 of the dose-adjustment period.

For Cohort III, PK assessments of carisbamate, S-enantiomer and its R-enantiomer plasma concentrations will be conducted on Days 1, 2 and 3 of the single dose period at pre dose and 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours after dosing and on Day 17 of the multiple-dose period at pre-dose and 2 hours after dosing; trough samples will be collected on Days 45 and 73 of the dose-adjustment period.

For Cohort IV, a sparse PK sampling approach will be used, and the time of PK sampling time will be based on the PK results from the other cohorts. A maximum of 2 to 4 time points on each day (1 and 17) will be collected.

Safety assessments include adverse event (AE) and concomitant medication reporting, clinical laboratory testing, vital sign measurements, 12 lead electrocardiograms (ECGs), physical examinations, and neurologic examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of LGS as evidenced by the following:

   1. More than 1 type of generalized seizure, including drop seizures (atonic, tonic, or myoclonic), for ≥6 months before Visit 1
   2. Previous electroencephalogram reporting diagnostic criteria for LGS (abnormal background activity accompanied by slow spike-and-wave pattern <2.5 Hz)
2. Male or female aged ≥2 years at the time of consent
3. Aged <11 years at the onset of LGS
4. Written informed consent signed by the subject or legal guardian prior to entering the study in accordance with the ICH GCP guidelines. Age appropriate assent will be obtained for children and adolescents. If the written informed consent is provided by the legal guardian because the subject is unable to do so, a written or verbal assent from the subject must also be obtained.
5. Receiving 1 to 3 concomitant AEDs at a stable dose for ≥30 days before Visit 1 (vagal nerve stimulation [VNS] and ketogenic diet, stable and ongoing for ≥30 days before Visit 1, do not count as AEDs)
6. In the Investigator's opinion, parents or caregivers must be able to report accurate seizure assessments during the screening and study periods and subjects must be able to ingest study drug
7. Body weight ≥8 kg for subjects enrolled in Cohort IV
8. Subjects with an implanted vagal nerve stimulator will be allowed if the vagal nerve stimulator was implanted at least 5 months prior to Visit 1 (Screening) and the stimulator parameters are not changed for 30 days prior to Visit 1 and for the duration of the study
9. Subjects following a ketogenic diet will be allowed as long as the diet has been stable for at least 30 days prior to Visit 1 (Screening) and will remain stable for the duration of the study.

Exclusion Criteria:

1. Progressive neurological disease
2. Prior treatment with carisbamate
3. Evidence of clinically significant disease or any medical condition that would compromise the subject's ability to safely complete the study
4. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the investigational medicine product
5. Acute disease state (e.g., nausea, vomiting, fever, or diarrhea) within 7 days before Day 1
6. Scheduled for surgery during the study
7. Ketogenic diet or VNS, unless stable and ongoing for ≥30 days before Visit 1
8. Treatment with an investigational drug or device ≥30 days before Visit 1
9. Status epilepticus within 12 weeks of Visit 1
10. Felbamate for <1 year (subjects taking felbamate for ≥1 year must have a stable dose for 60 days before Visit 1)
11. Concomitant use of vigabatrin or other medications known to be inducers of CYP3A
12. Use of drugs known as UGT inducers, e.g., carbamazepine, phenytoin, phenobarbital, primidone, or oxcarbazepine
13. Use of cannabinoids (any form), cannabidiols, or medical or recreational marijuana
14. Use of any prescription or non-prescription drugs, including over-the-counter medication, non-routine vitamins and herbal products within 2 weeks prior to study drug administration unless discussed and agreed with the Sponsor's medical representative in writing. (Medication used to treat TEAEs does not lead to a compulsory exclusion of subjects.)
15. Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours before Day 1 and until the end of each PK sampling period
16. Consumption of grapefruit or grapefruit-containing products within 72 hours before Day 1 and until the end of each PK sampling period
17. History of any serious drug-induced hypersensitivity reaction (including but not limited to Stevens Johnson syndrome, toxic epidermal necrolysis, Drug Rash with Eosinophilia and Systemic Symptoms [DRESS]) or any drug-related rash requiring hospitalization
18. History of AED-associated rash that involved conjunctiva or mucosae
19. History of more than one non-serious drug-related hypersensitivity reaction that required discontinuation of the medication
20. Significant clinical laboratory abnormalities, including elevation of serum AST or ALT more than 1.5 times ULN for age group, or any elevation of bilirubin or creatinine about the ULN for age group at Screening
21. Any clinically-significant uncontrolled medical illness, including hepatic or renal failure, ischemic disease, human immunodeficiency virus (HIV) infection, active sexually-transmitted disease (STD), active viral hepatitis, malignancy, or any disorder that in the judgement of the investigator places the subject at risk by participation in this study
22. History of drug-induced liver injury
23. Positive urine screen of drugs of abuse (if not due to concomitant medication, e.g. benzodiazepines as hypnotics) for adult and adolescent subjects.
24. Adrenocorticotropic hormone within the 6 months before Visit 1
25. History of anoxic episodes requiring resuscitation within 6 months before Visit 1, drug or alcohol dependency or abuse within approximately the last 2 years, or use of illegal recreational drugs
26. Females who are breastfeeding or pregnant at Screening or Baseline or who are of reproductive age and do not agree to be abstinent or to use highly effective contraception
27. Intermittent use of benzodiazepine of >4 single administrations in the month before Visit 1
28. Clinically significant abnormality on the 12-lead ECG at Screening, and any child or adolescent with a QTcF less than 330 ms or greater than 450 ms
29. Congenital short QT syndrome
30. Hypersensitivity to the study drug or any of the excipients
31. Psychotic disorder(s) or unstable recurrent affective disorder(s)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
The area under the curve (AUC) of carisbamate after a single and multiple doses of carisbamate. | Days 1-3, Day 17
  Safety Assessment
The maximum plasma concentration (Cmax) after a single and multiple doses of carisbamate. | Days 1-3, Day 17
  Safety assessment

SECONDARY OUTCOMES:
Safety - adverse events (AEs) reporting after a single and multiple doses of carisbamate. | Days 1-87
  Adverse event assessment for seriousness (yes, no), severity (mild, moderate, severe), affect on carisbamate dosing (increase, reduced, interrupted, withdrawn, no change), and outcome (recovered/resolved,recovered/resolved with sequelae, recovering/resolving, not recovered/not resolved, fatal or unknown).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, MD, Study Director — SK Life Science, Inc.
Locations (7):
- United States (7):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Duke Health, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Utah School of Medicine - Primary Children's Hospital (Primary Children's Medical Center), Salt Lake City, Utah
  - UW Valley Medical Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No